CLINICAL TRIAL: NCT05865509
Title: Comparison of the Escape Room and Storytelling Methods in Learning the Stress Response: A Randomized Controlled Study
Brief Title: Comparison of the Escape Room and Storytelling Methods in Learning the Stress Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Collaborators: Atılım University (Other)
Responsible Party: Principal Investigator, Nilgun Dogu, Asst. Prof., Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20221312
Record Dates: First submitted 2023-04-06; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Stress Response
Keywords: Escape room; Storytelling; Nursing; Game-based learning
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Escape room (Experimental): This group received training on stress response using the escape room method.
  Interventions: Other: Escape room
- Storytelling (Experimental): This group received training on stress response using the storytelling method.
  Interventions: Other: Storytelling

INTERVENTIONS:
Other: Escape room — Students were given training on stress response using the escape room method.
  Arms: Escape room
Other: Storytelling — Students were given training on stress response using the storytelling method.
  Arms: Storytelling

SUMMARY:
The goal of this randomised controlled study is to evaluate the effects of storytelling and escape room methods on the level of learning about stress response of nursing students and students' opinions about these methods.

The main questions it aims to answer are:

* Is there a difference between the pretest-posttest scores of the students who received training on stress response with the escape room method?
* Is there a difference between the pretest-posttest scores of the students who were trained on the stress response with the storytelling method?
* Is the difference between the knowledge levels of the students who received stress response training with the escape room and storytelling methods statistically significant? The students, who received training on stressors, stress response and the long-term effects of stress through lecture, were divided into two groups four weeks after this training and were retrained on the same subject with escape room and storytelling methods. Before and after the Escape room and storytelling practices, the students' knowledge of the stress response was evaluated. After both applications, focus group discussions were held with the students and their opinions and feedbacks on the applications were evaluated.

ELIGIBILITY:
Inclusion Criteria:

Nursing students taking internal medicine course

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Knowledge levels of students about stress response before the application. | On intervention day, just before application
  The knowledge level of the students about the stress response was evaluated by means of a form developed by the researchers after reviewing the literature. Students' Knowledge Assessing Form about the Stress Response, consisting of ten questions. The questions in the Students' Knowledge Assessing Form about the Stress Response were evaluated by a total of nine experts according to the Davis technique in terms of comprehensibility and content validity, and the content validity was found to be 1 (>0.80). Results from the Students' Knowledge Assessing Form about the Stress Response were evaluated based on the number of correct answers.
Knowledge levels of students about stress response after the application | On intervention day, immediately after application
  After the application, the knowledge levels of the students about stress response re-evaluated with the "Students' Knowledge Assessing Form about the Stress Response". After the application, the knowledge levels of the students about stress response re-evaluated with the "Students' Knowledge Assessing Form about the Stress Response". The difference between the knowledge levels of the students in the Escape room and Storytelling groups before and after the application was statistically evaluated using Mann Whitney U and Wilcoxon tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Nilgün Doğu, Ankara, Turkey (Türkiye)